CLINICAL TRIAL: NCT04176887
Title: Levetiracetam Versus Phenytoin in Management of Pediatric Status Epilepticus: a Randomized Clinical Trial
Brief Title: Levetiracetam Versus Phenytoin in Management of Pediatric Status Epilepticus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amira Hamed Darwish, Professor of pediatrics and Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUjune2018
Record Dates: First submitted 2019-09-11; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Comparison; the Efficacy of Levetireacetam; Phenytoin; Management of Pediatric Status Epilepticus
Keywords: Levetireacetam; Phenytoin; status epilepticus; children
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam; Phenytoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam (Experimental): The levetiracetam dose is 20- 40 mg/kg by intravenous infusion over 15 minute, a rate of 2-5 mg/kg/minute diluted in 100 ml with 0.9% sodium chloride as a single dose.
  Interventions: Drug: Levetiracetam Injection
- Phenytoin (Active Comparator): Phenytoin dose is 20-40 mg/kg/min by intravenous infusion over 30 minute, diluted with 0.9% sodium chloride to a maximum concentration of 10 mg/ml.
  Interventions: Drug: Phenytoin Injection

INTERVENTIONS:
Drug: Levetiracetam Injection — The levetiracetam dose is 20- 40 mg/kg by intravenous infusion over 15 minute, a rate of 2-5 mg/kg/minute diluted in 100 ml with 0.9% sodium chloride as a single dose.
  Other Names: levetiracetam
  Arms: Levetiracetam
Drug: Phenytoin Injection — Phenytoin dose is 20-40 mg/kg/min by intravenous infusion over 30 minute, diluted with 0.9% sodium chloride to a maximum concentration of 10 mg/ml.
  Other Names: Phenytoin
  Arms: Phenytoin

SUMMARY:
The study will be conducted on 60 children suffering from status epilepticus who will be admitted to Pediatric Neurology Unit and Pediatric ICU of Tanta Hospital University.

DETAILED DESCRIPTION:
The aim of this work is to compare the efficacy of Levetireacetam and Phenytoin in management of pediatric status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

* Children suffering from convulsive generalized tonic clonic status epilepticus at any age.

Exclusion Criteria:

* Non convulsive status epilepticus.
* Children with known contraindication or allergy to levetireacetam or phenytoin.

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
cessation of convulsion | 30 minutes
  seizure control based on stoppage of tonic and clonic movements and absence of epileptic activity in EEG

SECONDARY OUTCOMES:
bradycardia | 6 hours
  monitoring of heart rate
respiratory depression | 6 hours
  monitoring of respiratory rate
decreased conscious level | 6 hours
  Glasgow Coma Score
hypotension | 6 hours
  measurement of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Amira Darwish, MD, Principal Investigator — Tanta University Hospital
Locations (1):
- Tanta University, Faculty of Medicine, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided